CLINICAL TRIAL: NCT00721929
Title: Lipid-poor Adrenal Masses: Evaluation With Chemical Shift MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Gisela Mueller, MD, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2003-0148
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Adrenal Gland Disease
Keywords: adrenal glands, adrenal masses
MeSH Terms: conditions — Adrenal Gland Diseases

ARMS (1):
- adrenal mass group (Experimental)
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI — Magnetic Resonance Imaging

SUMMARY:
The purpose of this study is to determine if certain MRI sequences can accurately diagnose adrenal masses of unknown origin.

ELIGIBILITY:
Inclusion Criteria:

* Patients can participate in this study if they are 18 years of age or older and if they have had a Cat Scan (CT scan) performed with and without contrast media (medication given intravenously to enhance the CT images) or if patients are scheduled to have a CT scan performed and if the reason their physician ordered the CT is because they have an adrenal mass of an unknown type.

Exclusion Criteria:

* Patients, who have electrically, magnetically or mechanically activated implants such as heart pacemaker, magnetic surgical clips, prostheses or implanted neurological stimulator.
* Pregnant patients or patients who are lactating.
* A patient who is claustrophobic and would require sedation to complete the MRI exam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-10; Primary Completion 2010-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Diagnosis of either benign or malignant adrenal mass on pathology | 0-6 months
  definitive diagnosis of adrenal mass

SECONDARY OUTCOMES:
stability of growth of mass on follow up imaging | 3-24 months
  evidence for benign or malignant mass based on assessment of stability or growth

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States